CLINICAL TRIAL: NCT04116489
Title: Wildlife and Wellbeing: An Animal-Assisted Intervention for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Donna Perry, Associate Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H00016795; 1R21HD097771 (NIH)
Record Dates: First submitted 2019-07-22; First posted 2019-10-04 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wildlife Immersion Activity (Experimental): We will use a single group/ modified crossover design in which each participant receives an introductory forest walk followed by 3 wildlife immersion activity experiences in different settings .
  Interventions: Other: Forest walk; Other: Wildlife rehabilitation; Other: Wildlife sanctuary observation; Other: Bird feeding and watching

INTERVENTIONS:
Other: Forest walk — Participants will be provided with an educational program about the forest and take a guided forest walk.
Other: Wildlife rehabilitation — Participants will be provided with education on wildlife rehabilitation and assist with wildlife care such as feeding baby animals.
Other: Wildlife sanctuary observation — Participants will be provided an educational program on wildlife care and accompany park game keepers during animal feeding and will observe iconic wildlife.
Other: Bird feeding and watching — Participants will learn about bird identification and safe bird feeding. Bird feeders will be provided at the Soldier On facility for home bird feeding after study conclusion.

SUMMARY:
This study investigates a novel approach to animal-assisted interventions through a series of wildlife immersion activities (wildlife observation, wildlife rehabilitation and bird feeding/watching) for veterans who have suffered trauma as part of their military duty. Findings from this study will advance scientific knowledge about the benefits of wildlife activities for veterans with PTSD including the acceptability, feasibility, safety and preliminary influence on physical and mental well-being. The findings will be instrumental in advancing a new area of health intervention research for veterans in settings that are publicly accessible and family-oriented for sustainable, low-cost interventions with potential application in other populations.

DETAILED DESCRIPTION:
This study utilized a single group/ modified crossover design. The intervention included an introductory forest walk followed by 3 wildlife immersion activity experiences in different settings that offered different ways to experience wildlife. This included an introductory forest walk, a wildlife rehabilitation center, a wildlife sanctuary and a bird watching program. Each activity was conducted twice to minimize potential anxiety and novelty effects. Activities were conducted in small groups to provide peer support.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with PTSD/PTSD symptoms (per self report)
* Fully vaccinated against Covid-19, which is defined by the CDC as:

  * 2 weeks after second dose in a 2-dose series, such as the Pfizer or Moderna vaccines, or
  * 2 weeks after a single-dose vaccine, such as Johnson & Johnson's Janssen vaccine
* Age 18-70
* Comfortable interacting with animals
* Sufficient mobility to walk or navigate wheelchair up to one mile at leisurely pace
* Cognitive ability to complete assessments
* Service/ support animals are permitted as long as they meet the following criteria: the animal must be leashed, housebroken and with sufficient training that the owner has control over its barking and any other behaviors that would threaten the safety of other visitors or animals.
* Participants with visual or hearing impairments must have corrected vision and hearing through glasses and/ or hearing aid(s).
* No active addiction or intoxication as determined by 30 days or more free from drugs or alcohol abuse
* Willing to refrain from alcohol and illicit substances before and during activities
* No severe immunosuppression or other conditions with advisement by health care provider to limit or prevent contact with animals and birds
* No severe outdoor allergy.
* Not currently enrolled in the Veteran's Treatment Court program

Exclusion Criteria:

* Veterans without PTSD/PTSD symptoms (per self report
* Not fully vaccinated against Covid-19
* Age <18 or >70
* Not comfortable interacting with animals
* Not sufficiently mobile to walk or navigate wheelchair up to one mile at leisurely pace
* Cognitively unable to complete assessments
* Service/ support animals that do not meet the following criteria: leashed, housebroken and with sufficient training that the owner has control over its barking and any other behaviors that would threaten the safety of other visitors or animals.
* Participants with visual or hearing impairments who do not have corrected vision and hearing through glasses and/ or hearing aid(s).
* Active addiction or intoxication as determined by < 30 days free from drugs or alcohol abuse
* Not willing to refrain from alcohol and illicit substances before and during activities
* Severe immunosuppression or other conditions with advisement by health care provider to limit or prevent contact with animals and birds
* Severe outdoor allergy
* Currently enrolled in the Veteran's Treatment Court program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna J Perry, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wildlife Immersion Activity: We utilized a crossover design in which each participant received an introductory forest walk followed by 3 wildlife immersion activity experiences in different settings. Each activity was provided twice. Participants participated in each activity in the same order: Forest walk first, then wildlife rehabilitation, then wildlife sanctuary, then bird watching. There were not separate treatment arms.
  Forest walk: Participants were provided with an educational program about the forest and took a guided forest walk.
  Wildlife rehabilitation: Participants were provided with education on wildlife rehabilitation and assisted with wildlife care such as feeding baby animals.
  Wildlife sanctuary observation: Participants were provided an educational program on wildlife care and accompanied park game keepers during animal feeding and observation of wildlife.
  Bird feeding and watching: Participants will learn about bird identification and safe bird feeding. Bird feeders will be provided at the Soldier On facility for home bird feeding after study conclusion.
Period: Overall Study
Arm/Group | Wildlife Immersion Activity
Started | 19
Completed | 14
Not Completed | 5
Not completed — Participant left facility and was no longer eligible | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Veterans with PTSD
Groups:
- Wildlife Immersion Activity: We utilized a modified crossover design in which each participant received an introductory forest walk followed by 3 wildlife immersion activity experiences in different settings. Each activity was completed twice. All participants completed the activities in the same order: Forest walk first, then wildlife rehab, then wildlife sanctuary, then bird watching.
  Forest walk: Participants were provided with an educational program about the forest and undertook a guided forest walk.
  Wildlife rehabilitation: Participants were provided with education on wildlife rehabilitation and assisted with wildlife care such as feeding baby animals.
  Wildlife sanctuary observation: Participants were provided an educational program on wildlife care and observed animal care/ enrichment
  Bird feeding and watching: Participants were provided with education about bird characteristics and safe bird feeding. Bird feeders were provided for home bird feeding after study conclusion.
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Study participants [Number; unit: participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Recruitment of Study Participants
Description: Recruitment of study participants will be measured in order to determine the feasibility of delivering a wildlife program to veterans with PTSD.
Time Frame: at recruitment, day 1
Population: 28 participants that were screened were eligible for the study. 19 of these enrolled.
Measure: Number; unit: participants
Groups:
- Wildlife Immersion Activity: We will use a crossover design in which each participant receives an introductory forest walk followed by 3 wildlife immersion activity experiences in different settings .
  Forest walk: Participants will be provided with an educational program about the forest and take a guided forest walk.
  Wildlife rehabilitation: Participants will be provided with education on wildlife rehabilitation and assist with wildlife care such as feeding baby animals.
  Wildlife sanctuary observation: Participants will be provided an educational program on wildlife care and accompany park game keepers during animal feeding and will observe iconic wildlife.
  Bird feeding and watching: Participants will learn about bird identification and safe bird feeding. Bird feeders will be provided at the Soldier On facility for home bird feeding after study conclusion.
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 28
participants | 19

2. Primary Outcome: Change in Post Traumatic Stress Disorder (PTSD) Symptoms
Description: PTSD symptoms will be measured with the Posttraumatic Stress Disorder Checklist (PCL-5) which is a 20-item measure that assesses PTSD symptoms. Scores range from 0-80 with 33 or higher suggesting a provisional PTSD diagnosis. A higher score is worse.
Time Frame: Baseline to study conclusion (approximately 12 weeks per participant).
Population: All participants completed the baseline PCL-5 but only participants who finished the study completed the follow-up measure because the follow up survey was administered after the final activity.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 14
score on a scale | -6.56 (9.97)
Statistical Analysis 1: Comparison: Wildlife Immersion Activity; Test type: Superiority; p = .5272, Regression, Linear

3. Primary Outcome: Change in Perception of Well Being
Description: Perception of well being will be measured with the Warwick Edinburgh Mental Well Being Scale which is a 14 item instrument with scores ranging from 14 to 70. Higher scores indicate higher perceived well being.
Time Frame: Baseline to study conclusion (approximately 12 weeks per participant).
Population: Well being analysis included all participants and was adjusted for # of sessions attended.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 19
score on a scale | 3.17 (2.19)
Statistical Analysis 1: Comparison: Wildlife Immersion Activity; Test type: Superiority; p = .1657, Regression, Linear

4. Primary Outcome: Change in Depression
Description: Participant depression will be measured by the Center for the Epidemiological Study of Depression short form (CES-D-10) a 10 item instrument with a score range of 0-30 with higher scores indicating higher level of depression
Time Frame: Baseline to study conclusion (approximately 12 weeks per participant).
Population: Depression analysis included all participants and was adjusted for # of sessions attended.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 19
score on a scale | -1.84 (1.52)
Statistical Analysis 1: Comparison: Wildlife Immersion Activity; Test type: Superiority; p = .2437, Regression, Linear

5. Primary Outcome: Change in Level of Anxiety
Description: Anxiety will be measured by the Speilberger State/Trait Anxiety Inventory 6-item scale. Range is 20-80 with higher score being worse.
Time Frame: Baseline to after final activity (approximately 12 weeks per participant)
Population: Anxiety analysis included all participants and was adjusted for # of sessions attended.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 19
score on a scale | -7.72 (3.42)
Statistical Analysis 1: Comparison: Wildlife Immersion Activity; Test type: Other; p = .0373, Regression, Linear

6. Primary Outcome: Retention of Participants
Description: Number of participants who complete the study in comparison to those who enrolled in study (19)
Time Frame: Approximately 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Wildlife Immersion Activity
Number analyzed (Participants) | 19
Participants | 14

ADVERSE EVENTS:
Time Frame: Baseline to study conclusion, up to approximately 12 weeks per participant.
Description: Number of participants at risk is derived from # that attended each particular activity.
Groups:
- Forest Walk: Forest walk: Participants were provided with an educational program about the forest and took a guided forest walk.
- Wildlife Rehabilitation: Wildlife rehabilitation: Participants were provided with education on wildlife rehabilitation and assisted with wildlife care such as feeding baby animals.
- Wildlife Sanctuary Observation: Wildlife sanctuary observation: Participants were provided an educational program on wildlife care and accompanied park game keepers during animal feeding and observation of wildlife.
Arm/Group | Forest Walk | Wildlife Rehabilitation | Wildlife Sanctuary Observation | Bird Feeding and Watching
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/18 | 1/18 | 0/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forest Walk (N=18) | Wildlife Rehabilitation (N=18) | Wildlife Sanctuary Observation (N=13) | Bird Feeding and Watching (N=13)
Tick on skin (not embedded) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Occurred during Activity 1/ Forest Walk
Mild hypoglycemic symptoms during walk (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Occurred during Activity 1/ Forest Walk
Skin scratch from holding baby squirrel (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Occurred during Activity 2/ Wildlife rehabilitation care
Transient pain from acorn falling on shoulder (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Occurred during Activity 1/ Forest Walk

LIMITATIONS AND CAVEATS:
This study was limited by the need to put recruitment and intervention on hold for 1.5 years due to Covid, limiting the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04116489/Prot_SAP_000.pdf